CLINICAL TRIAL: NCT02544113
Title: A Randomized Controlled Clinical Trial of Thymoglobulin® and Extended Delay of Calcineurin Inhibitor Therapy for Renal Protection After Liver Transplantation. A Multi-Center Study
Brief Title: A Randomized Controlled Clinical Trial of Thymoglobulin® After Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Bijan Eghtesad, MD, Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-943
Record Dates: First submitted 2015-09-01; First posted 2015-09-09 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure | interventions — thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thymo (Experimental): Subjects randomized to the (Delay CNI) group will be treated with Thymoglobulin® (total dose of 4.5 mg/kg) administered in three doses; (each dose being 1.5 mg/kg - administered Day 0 [after transplant], Day 2, and Day 4 post transplant), along with CNI delay for 10 days. CNI will be initiated on postoperative (post-transplant) Day 10. Subjects will also receive a maintenance immunosuppression regimen of corticosteroids and MMF in accordance with the standard practice at each clinical center.
  Interventions: Drug: Thymoglobulin
- Control (Placebo Comparator): Subjects randomized to the (Early CNI) group (Control group) will receive no antibody therapy for induction and will start CNI therapy on postoperative (post-transplant) Day 2. Subjects will also receive a maintenance immunosuppression regimen of corticosteroids and MMF in accordance with the standard practice at each clinical center.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thymoglobulin — Treatment with thymoglobulin and delayed CNI post OLT
  Other Names: Anti-thymocyte Globulin
  Arms: Thymo
Drug: Placebo — Normal transplant immunosuppression
  Arms: Control

SUMMARY:
This is a 24-month, Phase II, multi-center, two-arm, randomized controlled study of adult patients receiving a single organ liver transplant from a deceased donor; the purpose being to determine the efficacy of Thymoglobulin® induction and delayed initiation of CNI in the long-term preservation of renal function after liver transplantation. This study is based on the outcomes of an earlier phase 1 pilot study which was performed at the Cleveland Clinic.

This study will be conducted at 3 centers, with 110 subjects randomized 1:1 into two groups: Group 1 will receive Thymoglobulin® induction, (4.5 mg/Kg, in 3 doses of 1.5 mg/Kg/dose) with delayed initiation of CNI to begin on Day 10 post LT. Group 2 will receive early CNI initiation (to be started no later than Day 2 post LT), and no Thymoglobulin® induction (or any other antibody).

All subjects will also receive a maintenance immunosuppressive regimen consisting of corticosteroids and mycophenolate mofetil (MMF) according to standard of practice in orthotopic liver transplantation (OLT).

Subjects will be consented pre-transplant. Participation may last up to 12 months post OLT. There are 15 study-related visits which will be completed during standard of care (SOC) visits.

DETAILED DESCRIPTION:
Functional recovery of renal function from acute renal failure occurs in 75% of patients at approximately 14 days after onset of the disease. In liver transplantation, intraoperative hemodynamic insults typically lead to acute renal failure which may be further worsened by exposure to CNI therapy in the early postoperative period. In practice, patients who demonstrate early evidence of acute renal failure often have their CNI therapy delayed for 4-5 days. This duration of CNI delay is too short to have any salutary effect on the course or severity of acute kidney injury as less than 20% of patients experience any functional recovery by day 5.

Thymoglobulin® (Sanofi, Cambridge, MA) is a polyclonal immunosuppressive agent that is derived from rabbits immunized with pediatric thymocytes. It contains antibodies to a wide variety of T-cell antigens and major histocompatibility complex (MHC) antigens and is approved for the treatment of kidney rejection by the FDA. Thymoglobulin® has been shown to be a safe and efficacious induction therapy that permits delayed exposure to CNI therapy while preventing the occurrence of acute rejection in kidney transplantation. The investigators hypothesize that any perioperative insult leading to AKI in OLT recipients is unlikely to be beneficially impacted by a short delay of CNI introduction. Further hypothesized is that avoidance of CNI for 10 days will have a beneficial effect on the course and severity of perioperative AKI. Since perioperative AKI is a potent risk factor for chronic kidney disease (CKD) in the late post-transplant period, also hypothesized is that minimizing the risk and severity of AKI with prolonged delayed exposure to CNI will have a beneficial effect on renal function late after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing deceased donor solitary liver transplantation
* Age 18-75 years at the time of transplantation
* Willingness and ability to comply with the study procedures
* Signed informed consent form
* For patients with Hepatocellular carcinoma as indication for OLT, (must be within the Milan Criteria)
* Hepatitis C, positive or negative, patients

Exclusion Criteria:

* Prior kidney transplantation
* Congenital or iatrogenic absence of one kidney
* Subjects on renal replacement therapy at the time of OLT
* MELD score >34
* HIV positive patient
* Patient with current severe systemic infection
* History of bacterial peritonitis within 30 days prior to OLT
* Active infection or recent infection within 30 days prior to OLT
* Use of a calcineurin inhibitor continuously for more than 90 days within the past 6 months
* History of hypersensitivity to Thymoglobulin®, rabbits or tacrolimus
* Pregnant and/or nursing (lactating) females.
* Women of childbearing age who are unwilling to use effective contraception during the duration of the study, and for 30 days after study participation and/or last dose of Study Drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-12; Primary Completion 2018-06-26 (Actual); Study Completion 2020-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Eghtesad, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - Cleveland Clinic Florida, Weston, Florida
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Cleveland Clinic (Main Campus), Cleveland, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Nair A, Coromina Hernandez L, Shah S, Zervos X, Zimmerman M, Sasaki K, Diago T, Hashimoto K, Fujiki M, Aucejo F, Bollinger J, Kaiser TL, Miller CM, Quintini C, Fung JJ, Eghtesad B. Induction Therapy With Antithymocyte Globulin and Delayed Calcineurin Inhibitor Initiation for Renal Protection in Liver Transplantation: A Multicenter Randomized Controlled Phase II-B Trial. Transplantation. 2022 May 1;106(5):997-1003. doi: 10.1097/TP.0000000000003904. Epub 2021 Jul 27. PMID 34319926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thymo | Control
Started | 55 | 55
Completed | 52 | 51
Not Completed | 3 | 4
Not completed — Death | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymo | Control | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.2) | 59.8 (12.1) | 58.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 40 | 33 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 52 | 49 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Acute Kidney Injury (AKI) as Assessed by Change in Serum Creatinine From Baseline to 30 Days Post-transplant
Description: Change in serum creatinine from baseline to 30 days post-transplant. Higher values are associated with worse outcomes, and values greater than 0.3 mg/dL are suggestive of acute kidney injury.
Time Frame: 30 days post-transplant
Population: Analysis was performed on a complete-case basis. Outcome measure data was not available for all enrolled subjects.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Thymo | Control
Number analyzed (Participants) | 43 | 52
mg/dL | .01 (0.53) | .06 (0.28)

2. Secondary Outcome: Number of Participants Experiencing Acute Cellular Rejection
Description: The number of participants experiencing acute cellular rejection, as determined by biopsy.
Time Frame: 30 days post OLT
Measure: Count of Participants; unit: Participants
Arm/Group | Thymo | Control
Number analyzed (Participants) | 55 | 55
Participants | 9 | 7

3. Secondary Outcome: Graft Survival
Description: Number of participants who did not require retransplantation
Time Frame: 6 months post OLT
Measure: Count of Participants; unit: Participants
Arm/Group | Thymo | Control
Number analyzed (Participants) | 55 | 55
Participants | 55 | 55

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 12 months
Description: Participants were assessed for adverse events at regular study visits
Arm/Group | Thymo | Control
All-Cause Mortality (participants affected / at risk) | 3/55 | 4/55
Serious Adverse Events (participants affected / at risk) | 13/55 | 13/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymo (N=55) | Control (N=55)
Infection (Infections and infestations) | 8 (9) | 8 (11)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Hypertension (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Hepatic Artery Thrombosis (Hepatobiliary disorders) | 1 (3) | 1 (1)
Portal Vein Stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal Liver Function Tests (Hepatobiliary disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT02544113/Prot_SAP_000.pdf